CLINICAL TRIAL: NCT01479023
Title: A Phase 1 Evaluation of 64Cu-DOTA-U3-1287 in Subjects With Advanced Solid Tumors and Determination of Tumor Receptor Occupancy by U3-1287
Brief Title: Evaluation of 64Cu-DOTA-U3-1287 in Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: treatment was not working
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201202074
Record Dates: First submitted 2011-11-17; First posted 2011-11-24 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Carcinoma; Sarcoma; Lymphoma
MeSH Terms: conditions — Carcinoma; Sarcoma; Lymphoma | interventions — patritumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Cohort 1 (Experimental): 64Cu-DOTA-U3-1287 at a radiotracer dosage of 8-15 mCI and ≤ 0.2 mg of DOTA-U3-1287 on Day 1.
  Patient will have option to continue to Part 2 (extension phase).
  Interventions: Drug: 64Cu-DOTA-U3-1287; Drug: U3-1287 (unlabeled)
- Cohort 2 (Experimental): 64Cu-DOTA-U3-1287 at the radiotracer dosage defined by Cohort 1 and ≤ 0.2 mg of DOTA-U3-1287 on Day 1.
  9.0 mg/kg unlabeled U3-1287 followed by a second dose of ≤ 0.2 mg 64Cu-DOTA-U3-1287 on Day 8.
  Patient will have option to continue to Part 2 (extension phase).
  Interventions: Drug: 64Cu-DOTA-U3-1287; Drug: U3-1287 (unlabeled)
- Cohort 3 (Experimental): 64Cu-DOTA-U3-1287 at the radiotracer dosage defined by Cohort 1 and ≤ 0.2 mg of DOTA-U3-1287 on Day 1.
  12.0 mg/kg unlabeled U3-1287 followed by a second dose of ≤ 0.2 mg 64Cu-DOTA-U3-1287 on Day 8.
  Patient will have option to continue to Part 2 (extension phase).
  Interventions: Drug: 64Cu-DOTA-U3-1287; Drug: U3-1287 (unlabeled)
- Cohort 3a (Experimental): 64Cu-DOTA-U3-1287 at the radiotracer dosage defined by Cohort 1 and ≤ 0.2 mg of DOTA-U3-1287 on Day 1.
  15.0 mg/kg unlabeled U3-1287 followed by a second dose of ≤ 0.2 mg 64Cu-DOTA-U3-1287 on Day 8.
  Patient will have option to continue to Part 2 (extension phase).
  Interventions: Drug: 64Cu-DOTA-U3-1287; Drug: U3-1287 (unlabeled)
- Cohort 4 (Experimental): 64Cu-DOTA-U3-1287 at the radiotracer dosage defined by Cohort 1 and ≤ 0.2 mg of DOTA-U3-1287 on Day 1.
  18.0 mg/kg unlabeled U3-1287 followed by a second dose of ≤ 0.2 mg 64Cu-DOTA-U3-1287 on Day 8.
  Patient will have option to continue to Part 2 (extension phase).
  Interventions: Drug: 64Cu-DOTA-U3-1287; Drug: U3-1287 (unlabeled)
- Cohort 5 (Experimental): 64Cu-DOTA-U3-1287 at the radiotracer dosage defined by Cohort 1 and ≤ 0.2 mg of DOTA-U3-1287 on Day 1.
  TBD (to be determined) mg/kg unlabeled U3-1287 followed by a second dose of ≤ 0.2 mg 64Cu-DOTA-U3-1287 on Day 8.
  Patient will have option to continue to Part 2 (extension phase).
  Interventions: Drug: 64Cu-DOTA-U3-1287; Drug: U3-1287 (unlabeled)
- Part 2 (extension phase) (Experimental): Loading dose of 18.0 mg/kg unlabeled U3-1287 followed by 9.0 mg/kg unlabeled U3-1287 every 3 weeks.
  Interventions: Drug: 64Cu-DOTA-U3-1287; Drug: U3-1287 (unlabeled)

INTERVENTIONS:
Drug: 64Cu-DOTA-U3-1287
Drug: U3-1287 (unlabeled)

SUMMARY:
2.1 Primary Objectives

1. To measure the human dosimetry of 64Cu-DOTA-U3-1287 in subjects with advanced solid tumors (Cohort 1 only)
2. To calculate HER3 receptor occupancy (via quantification of the tumor-localized PET signal produced by 64Cu-DOTA-U3-1287 in the absence and presence of competing unlabeled U3-1287 in subjects with advanced solid tumors (Cohorts 2 through 5))
3. To determine the safety and tolerability of 64Cu-DOTA-U3-1287 (all cohorts)

2.2 Secondary Objectives

1. To determine the relationship between U3-1287 serum concentration and HER3 receptor occupancy (as measured by PET/CT) in subjects with advanced solid tumors
2. To measure the tumor response rate as defined by Response Evaluation Criteria in Solid Tumors (RECIST 1.1) in subjects with advanced solid tumors treated with U3-1287 (Part 2 only)
3. To characterize the PK exposure of U3 1287 when administered intravenously to patients with advanced solid malignancies.
4. To measure the rate of anti-U3-1287 human antibody development in subjects with advanced solid tumors treated with U3 1287 monotherapy

2.3 Exploratory Objectives

1. To assess tumor volume changes after U3-1287 treatment by CT or magnetic resonance imaging (MRI) (Part 2 only)
2. To assess blood, body fluid/tissue, and tumor specimens for potential biomarkers (e.g., proteins and transcripts) that predict response to U3-1287
3. To obtain tumor samples for DNA extraction for analysis of potential predictors of response to U3-1287 and any related genes as suggested by emerging data

ELIGIBILITY:
Inclusion Criteria:

* Patient must have measurable disease as defined by RECIST 1.1, with the additional requirement of at least one lesion ≥ 1.5 cm on CT scan or detectable on FDG-PET performed within 30 days prior to screening
* Patient must have a tumor where HER3 expression is expected (this includes breast, colon, lung, prostate, ovarian, cervical, endometrial, gastric, pancreatic, bladder, head and neck, liver, and esophageal cancer, but other tumors will be considered based on emerging HER3 expression data)
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Patient must have pathologically documented, definitively diagnosed, advanced solid tumors that are refractory to standard treatment or for which no curative therapy is available
* Patient must have adequate hematologic and organ function as follows:

  * Absolute neutrophils count (ANC) ≥ 1.5 x 109/L
  * Platelet count ≥ 100 x 109/L
  * Hemoglobin ≥ 9 g/dL
  * Serum creatinine ≤ 2 x IULN
  * AST ≤ 2.5 x IULN (≤ 5.0 x IULN if attributable to liver metastasis)
  * ALT ≤ 2.5 x IULN (≤ 5.0 x IULN if attributable to liver metastasis)
  * Alkaline phosphatase ≤ 2.0 x ULN (if bone or liver metastases are present, < 5 x ULN)
  * Total bilirubin ≤ 1.5 IULN
  * Amylase or lipase ≤ 2.0 x IULN
  * Prothrombin time (PT) or partial thromboplastin time (PTT) ≤ 1.5 x IULN
* Patient must have an LVEF of ≥ 50%
* Patient must be ≥ 18 years old
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry, for the duration of study participation, and for 6 months following the completion of study treatment; should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Patient must be willing and able to undergo the imaging studies outlined in the protocol (in the opinion of the investigator)
* Patient must be able to understand and willing to sign an institutional review board (IRB) approved informed consent form
* Patient must have archival tissue available for HER3 expression analysis

Exclusion Criteria:

* Patient must not have the liver and/or spleen as the only site(s) of disease (as PET/CT imaging of 64Cu-DOTA-U3-1287 may be difficult in these anatomic locations)
* Patient must not have any unresolved toxicities > grade 1 with the exception of grade 2 lymphopenia and/or alopecia from prior anti-cancer therapy Note: Grade 2 or 3 toxicities from prior therapy that are considered irreversible (defined as having been present and stable for > 3 months), such as ifosfamide-related proteinuria, or treatment related neuropathy, may be allowed if they are not otherwise described in the exclusion criteria AND the PI and Daiichi Sankyo both agree that this patient may be included
* Patient must not have untreated or symptomatic primary central nervous system metastases or symptoms of brain metastases; any stereotactic radiation or whole brain radiation therapy must have been completed at least 4 weeks prior to study entry
* Patient must not have ascites or pleural effusion requiring medical intervention
* Patient must not have had a myocardial infarction within 6 months of Day 1 or any unstable or uncontrolled disease/condition related to or impacting cardiac function (i.e., unstable angina, congestive heart failure, New York Heart Association > class II, uncontrolled hypertension [diastolic > 95 mmHg; systolic >140 mmHg])
* Patient not have cardiac arrhythmia or clinically significant ECG abnormalities
* Patient must not be known to be positive for human immunodeficiency virus (HIV) infection, hepatitis C virus, or chronic active hepatitis B infection
* Patient must not have a known sensitivity to any components of the formulation
* Patient must not be receiving any concomitant antitumor treatment or chemotherapy, radiotherapy, and hormonal therapy (with the exception of Lupron for prostate cancer and SERMS for breast cancer subjects) within 4 weeks of Day 1 (6 weeks for nitrosoureas or mitomycin and 2 weeks for small molecule tyrosine kinase inhibitors)
* Patient must not be receiving any concomitant immunosuppressant therapy (cyclosporine A, FK506, etc., or chronic > 5 mg/d of prednisone)
* Patient must not be receiving any other concomitant investigational procedures and must not have participated in any other clinical trial with an investigational device or agent within 4 weeks of the first dose of 64Cu-DOTA-U3-1287
* Patient must not have had any previous exposure to U3-1287
* Patient must not have had any previous treatment with HER3 antagonists
* Patient must not have had G-CSF support therapy within 2 weeks of Day 1
* Patient must not have received red blood cell (RBC) transfusion within 2 weeks of Day 1
* Patient must not have received platelet transfusion within 2 weeks of Day 1
* Patient must not be pregnant or planning to become pregnant within 6 months after the end of treatment; patient must not be breastfeeding
* Patient must not have a known sensitivity to any of the products to be administered during dosing, including excipients, radiolabeled agents
* Patient must not have had major surgery within 28 days of Day 1 or predicted need for major surgery while on study
* Patient must not schedule any elective surgeries (with the exception of port placement or replacement) during his/her participation in the study and through 28 days after the last administration of U3-1287
* Patient must not have any comorbid medical disorder that may increase the risk of toxicity in the opinion of the investigator or sponsor
* Inclusion of Women and Minorities

Both men and women and members of all races and ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-04; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Human dosimetry of 64Cu-DOTA-U3-1287 in subjects with advanced solid tumors (Cohort 1 only) | 2 days
  Measurement of the human dosimetry at 3 hours post dose, 24 hours post dose and 48 hours post dose.
HER3 receptor occupancy (via quantification of the tumor-localized PET signal produced by 64Cu-DOTA-U3-1287 in the absence and presence of competing unlabeled U3-1287 in subjects with advanced solid tumors (Cohorts 2 through 5)) | 9 days
  Calculation of HER3 receptor occupancy (via quantification of the tumor-localized PET signal produced by 64Cu-DOTA-U3-1287 in the absence and presence of competing unlabeled U3-1287
Safety and tolerability of 64Cu-DOTA-U3-1287 (all cohorts) | From first receiving study treatment until the 8-week follow-up after the conclusion of treatment or death
  Based on adverse events according to NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0

SECONDARY OUTCOMES:
Relationship between U3-1287 serum concentration and HER3 receptor occupancy in subjects with advanced solid tumors | 9 days
  Measured by PET/CT at 24 hours post dose Day 1 and 24 hours post dose Day 8
Tumor response rate in subjects with advanced solid tumors treated with U3-1287 (Part 2 only) | Followed for 8 weeks following last administration of study or until death, whichever occurs first
  Defined by Response Evaluation Criteria in Solid Tumors (RECIST 1.1. Screening, after two dose (6 weeks) of U3-1287 during Part 2, and every 9 weeks thereafter.
PK exposure of U3-1287 when administered intravenously to patients with advanced solid malignancies. | Various timepoints depending on cohort
  Cohort 1 Part 1 = Day 1 predose, end of infusion, hour 3, 24 hours, 48 hours, and 72 hours.
  Cohort 1 Part 2 = Day 8 predose, 5 minutes pre-end of infusion, hour 6, day 9, day 15, day 22, and then every 3 weeks.
  Cohorts 2-5 Part 1 = Day 1 predose, end of infusion, 24 hours, Day 8 predose, end of infusion, and Day 9.
  Cohorts 2-5 Part 2 = Day 29 predose, end of infusion, Day 30, and every 3 weeks.
Rate of anti-U3-1287 human antibody development in subjects with advanced solid tumors treated with U3-1287 monotherapy | Up to 1 year from the last dose of study drug
  Pre-infusion on Day 1 of every cycle and end of study treatment visit.
  For patients positive for anti-U3-1287 neutralizing antibody on the serum sample drawn at the final visit, additional serum samples should be obtained until the level returns to baseline (or becomes negative) or up to 1 year from the last dose of study drug or if the patient starts another therapy for his/her cancer, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: A. Craig Lockhart, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Lockhart AC, Liu Y, Dehdashti F, Laforest R, Picus J, Frye J, Trull L, Belanger S, Desai M, Mahmood S, Mendell J, Welch MJ, Siegel BA. Phase 1 Evaluation of [(64)Cu]DOTA-Patritumab to Assess Dosimetry, Apparent Receptor Occupancy, and Safety in Subjects with Advanced Solid Tumors. Mol Imaging Biol. 2016 Jun;18(3):446-53. doi: 10.1007/s11307-015-0912-y. PMID 26567113
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu